CLINICAL TRIAL: NCT01699555
Title: Randomized Placebo-Controlled First-in-Human Study With GNbAC1
Brief Title: First-in-Human Study With GNbAC1 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GeNeuro Innovation SAS (Industry)
Responsible Party: Sponsor
Organization: GeNeuro SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GNC-001
Record Dates: First submitted 2012-09-27; First posted 2012-10-03 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2012-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; GNbAC1; Monoclonal antibody; Multiple Sclerosis Associated Retrovirus (MSRV); Temelimab
MeSH Terms: conditions — Multiple Sclerosis | interventions — temelimab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GNbAC1 (Experimental): Single dose intravenous (IV) GNbAC1 of 0.0025mg/kg, 0.025mg/kg, 0.15mg/kg, 0.60mg/kg, 2.00mg/kg or 6.00mg/kg
  Interventions: Biological: GNbAC1
- GNbAC1 placebo (Placebo Comparator): Single dose intravenous (IV) GNbAC1 placebo
  Interventions: Biological: GNbAC1 placebo

INTERVENTIONS:
Biological: GNbAC1 — Single dose intravenous (IV) GNbAC1 of 0.0025mg/kg, 0.025mg/kg, 0.15mg/kg, 0.60mg/kg, 2.00mg/kg or 6.00mg/kg
  Arms: GNbAC1
Biological: GNbAC1 placebo — Single dose intravenous (IV) GNbAC1 placebo
  Arms: GNbAC1 placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of single ascending doses of GNbAC1 in healthy male subjects.

DETAILED DESCRIPTION:
Scientific research has shown that the expression of genes of a virus which is integrated in the Human genetic material, the Multiple Sclerosis associated RetroVirus (MSRV) could play a critical role in the causation of multiple sclerosis. GNbAC1 is an experimental medication, which neutralizes (i.e. inactivates) a protein of MSRV that might contribute to the development or deterioration of multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Male healthy subjects, 18-55 years of age and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram and laboratory tests at Screening and confirmed at baseline.
* Clinically acceptable for the purposes of the study sitting blood pressure and pulse rate, i.e.: BP: 100 - 150 mm Hg systolic, 50 - 95 mm Hg diastolic and pulse rate: 45 - 100 bpm. Blood pressure and pulse will be measured after 3 minutes resting in a sitting position.
* Body mass index between 18.5 and 30.0 kg/m2 and body weight in the 50 - 95 kg range.
* No need for regular concomitant medication
* Subjects with partners of childbearing potential have to use adequate contraception during, and for at least the four weeks after administration of study medication. Adequate contraception is defined as usage by at least one of the partners of a barrier method of contraception, together with usage by the female partner, commencing at least three months prior to Screening, of a stable regimen of any form of hormonal contraception or an intra-uterine device. Use of abstinence alone is not considered adequate. Use of a barrier method alone is considered adequate only if the subject was vasectomized at least six months prior to Screening.
* Ability to communicate well with the investigator and comply with the requirements of the entire study.
* The subject has given written consent to participate in the study.

Exclusion Criteria:

* History of serious adverse reactions or hypersensitivity to any drug.
* Presence or history of any allergy requiring acute or chronic treatment (seasonal allergic rhinitis which requires no treatment may be tolerated).
* Abnormal physical findings of clinical significance at the Screening or baseline examination which would interfere with the objectives of the study.
* Need of any prescription medication within 30 days prior to the administration of the drug and/or nonprescription medication within 7 days prior to the administration of the drug or anticipated need for any concomitant medication during the study.
* Participation in a clinical trial during the previous 4 weeks, i.e. from completion of the previous trial to the planned first administration of the current trial.
* Loss of 500 mL blood or more during the 3 month period before the screening visit of the study, e.g. as a donor.
* Existence of any surgical or medical condition which might relevantly interfere with the subject safety, the distribution, metabolism or excretion of the drug or the study assessments, i.e. impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhea or conditions associated with total or partial obstruction of the urinary tract.
* Symptoms of a significant (upon Investigator's medical judgment) somatic or mental illness in the two week period preceding drug administration.
* History or clinical evidence of significant cardiovascular, respiratory, renal, hepatic,gastrointestinal, hematological, neurologic or other disease.
* History of hepatitis B and / or C and / or positive serology results which indicate the presence of hepatitis B and / or C.
* Positive results from the HIV serology.
* Positive for MSRV env by RNA PCR
* Clinically significant abnormal laboratory values (as determined by the Principal Investigator in consultation with the sponsor) at the Screening or baseline evaluation.
* History of serious mental disorders.
* History of alcohol or drug abuse in the last 3 years.
* Heavy smokers, i.e. more than 10 cigarettes per day and/or unwillingness to refrain from smoking during the entire in-house period.
* Positive results of the drug Screening.
* Need for a vaccination from Screening to End of Study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2011-07; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
number of reported adverse events for healthy male subjects receiving single ascending doses of GNbAC1. | 64 days
  the number of adverse events along with the results of physical examinations, ECG and clinical laboratory tests will be used to determine the safety profile of GNbAC1.

SECONDARY OUTCOMES:
pharmacokinetics (PK) characteristics following administration of single ascending doses of GNbAC1 in healthy male subjects | 64 days
  the following parameters will be determined: serum concentrations of GNbAC1 and the derived PK parameters AUC0-inf, AUC0-tlast, %AUC, Cmax, tmax, t1/2, λz, CL, Vss, Vz, MRT.
immunogenicity of GNbAC1 | 64 days

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Kamtchoua, M.D, Principal Investigator — Covance Clinical Research Unit AG

REFERENCES:
- [Result] Curtin F, Lang AB, Perron H, Laumonier M, Vidal V, Porchet HC, Hartung HP. GNbAC1, a humanized monoclonal antibody against the envelope protein of multiple sclerosis-associated endogenous retrovirus: a first-in-humans randomized clinical study. Clin Ther. 2012 Dec;34(12):2268-78. doi: 10.1016/j.clinthera.2012.11.006. Epub 2012 Nov 29. PMID 23200102